CLINICAL TRIAL: NCT06179758
Title: Remote MS Care in Antwerp
Acronym: ReMSCA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Janssen-Cilag div. of Johnson&Johnson SE (Industry); icometrix (Industry); Ziekenhuis Netwerk Antwerpen (ZNA) (Other); AZ Klina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 3258
Record Dates: First submitted 2023-10-03; First posted 2023-12-22 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-01

CONDITIONS: Multiple Sclerosis
Keywords: remote monitoring
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- open-label interventional arm (Experimental)
  Interventions: Device: icompanion app

INTERVENTIONS:
Device: icompanion app — use of the icompanion app as a digital telemonitoring solution

SUMMARY:
Current clinical follow-up of multiple sclerosis (MS) patients suffers from some challenges, as many patients indicate they want to take up a more active role in the decision-making process. However, more than half of MS patients do not consider themselves well informed about their disease. Communication between patients and healthcare professionals (HCPs) has also been reported to be suboptimal, with incorrect alignment between patients and HCPs as a result and relapses going undetected. Digital telemonitoring tools could play a role in educating MS patients, allowing them to take up a more active role in the clinical decision-making process. Additionally, remote monitoring could lead to a better alignment between patient and HCPs and could ultimately even lead to a more efficient clinical workflow.

In this study, the investigators will investigate an existing digital telemonitoring solution called icompanion, developed by Icometrix. icompanion is a class 1 medical device in US (Food and Drug Administration - FDA) and Europe (Medical Device Directive - MDD). Using the icompanion MS app and website, patients can keep a diary, log symptoms, and perform tests for body function, cognitive function and fatigue based on clinically validated patient-reported outcomes (PROs). In addition, MS patients can add treatment information, from disease modifying therapies (DMTs) to symptomatic and rehabilitation treatments, and set reminders on when to take or perform their treatment. Furthermore, patients can easily upload their magnetic resonance imaging (MRI) scans (via the patient website) and view them (via the patient website and app) as well as learn about topics related to MS (e.g., MS types, MRI lesions). Finally, patients can prepare their consultations using a pre-visit checklist, the answers of which are also shared with the patient's clinical team.

This study aims to evaluate the feasibility to use this app in a population of 100 MS patients in Antwerp, in three clinical centres. For this, the following objectives have been set forth:

* The primary objective is to evaluate the usability and acceptance of a digital remote monitoring solution for MS (icompanion).
* The secondary objectives are:

  1. To evaluate the relationship between MS patients' subjective health experience, disease control and disease acceptation (by using the Health Monitor) and adherence and usability
  2. To evaluate the impact of the use of the solution on the Health Monitor profile (reflecting patients' subjective health experience, disease control and disease acceptation) in a pre- versus post-intervention analysis
  3. To evaluate the impact of the solution on the MS patients' disease self-management, by use of the Multiple Sclerosis Self-Management Scale-Revised (MSSM-R)
  4. To evaluate the impact of the solution on the clinical visit workflow, by using visual analogue scales with custom questions about impact on workflow
* The tertiary objectives are:

  1. To evaluate the concordance between patient-reported and clinician-assessed values of some of the parameters collected by the icompanion default dataset (e.g., patient-reported Expanded Disability Status Scale (EDSS), daily steps), when available
  2. To evaluate the app features most used by patient users
  3. To evaluate the web portal features most used by HCP users

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of multiple sclerosis (MS, including relapsing-remitting MS, primary-progressive MS and secondary-progressive MS, in accordance with 2017 revisions of McDonald criteria and disease course definitions of Lublin,
2. Age 18 or above,
3. Able to give informed consent (written or verbal with witness signing on behalf of patient) and to adhere to study procedures,
4. Dutch/Flemish speaking.

Exclusion Criteria:

1. Unable or unwilling to use the smartphone-based icompanion app.
2. Prior use of the icompanion app.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
the acceptance of a digital remote monitoring solution for MS (icompanion) (adherence number) | month 2, month 6, month 12
  measurement variable: adherence number (adherence defined as use of the icompanion app minimally once a month, score between 0 and 100%)
the usability of a digital remote monitoring solution for MS (icompanion) | month 2, month 6, month 12 (for patients), clinical visit 1 and 2 (for health care professionals, visit 1 between three to six months following inclusion and visit 2 between six to twelve months following inclusion, depending on individual follow-up)
  measurement variable: system usability scale (10 questions, score between 10 and 50, with higher scores meaning a better usability)

SECONDARY OUTCOMES:
the correlation between MS patients' subjective health experience, disease control and disease acceptation (by using the Health Monitor) and adherence and usability | month 0, month 2, month 6, month 12
  the correlation between an individual's Health Monitor segment (4-segment segmentation approach based on a short questionnaire of 6 questions, reflecting an individual's sense of control and acceptance) and his/her adherence and estimation of the usability of the icompanion app (using the system usability scale (10 questions, score between 10 and 50, with higher scores meaning a better usability) will be assessed
the impact of the use of the solution on the Health Monitor profile (reflecting patients' subjective health experience, disease control and disease acceptation) in a pre- versus post-intervention analysis | month 0, month 2, month 6, month 12
  the evolution of an individual's Health Monitor segment (4-segment segmentation approach based on a short questionnaire of 6 questions, reflecting an individual's sense of control and acceptance) before and after use of the icompanion app
the impact of the use the solution on the MS patients' disease self-management, by use of the MSSM-R | month 0, month 2, month 6, month 12
  measurement variable: Multiple Sclerosis Self-Management Scale-Revised (MSSM-R, 24 questions, score between 24 and 120, with higher scores meaning a higher degree of disease self-management)
the impact of the solution on the clinical visit workflow, by using visual analogue scales with custom questions about impact on workflow | clinical visit 1 and 2 clinical visit 1 and 2 (for patients and health care professionals, visit 1 between three to six months following inclusion and visit 2 between six to twelve months following inclusion, depending on individual follow-up)
  measurement variable: visual analogue scales with custom questions about impact on clinical visit (5 questions, score between 5 and 25, with higher scores meaning a better impact on the clinical visit workflow)

OTHER OUTCOMES:
the concordance between patient-reported and clinician-assessed values of some of the parameters collected by the icompanion default dataset, when available | continuously throughout the study, for an estimated duration of 6 to 12 months
  measurement variable: icompanion dataset (e.g., patient-reported Expanded Disability Status Scale (EDSS), score from 0 to 10, with lower scores meaning less disease-related signs and symptoms)
the app features most used by patient users | continuously throughout the study, for an estimated duration of 6 to 12 months
  measurement variable: usage rate of the individual app features
the web portal features most used by health care professional users | continuously throughout the study, for an estimated duration of 6 to 12 months
  measurement variable: usage rate of the individual features of the icompanion web portal

CONTACTS AND LOCATIONS:
Locations (3):
- Belgium (3):
  - University Hospital Antwerp, Edegem, Antwerpen
  - ZAS Middelheim, Antwerp
  - AZ Klina, Brasschaat

IPD SHARING:
Plan to Share IPD: Undecided